CLINICAL TRIAL: NCT02467166
Title: A Prospective, Non-Randomized Study to Evaluate the CIRCA Esophageal Temperature Monitoring System in Prevention of Esophageal Lesions Following Atrial Fibrillation Radiofrequency Catheter Ablation
Brief Title: Evaluation of the CIRCA Monitoring System in Prevention of Esophageal Lesions Following RFCA
Acronym: CIRCA-EGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Circa Scientific, Inc. (Industry)
Responsible Party: Principal Investigator, Greg Feld, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 150018
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation
Keywords: esophagoscopy; atrial fibrillation ablation; radio frequency catheter ablation; esophageal lesion; arrhythmia; atrial fibrillation; AF; esophageal damage
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Circa™ Probe (Experimental): The Circa™ Probe will be used during the RFCA to monitor esophageal temperature. Following ablation, the esophagoscopy will be performed to examine the esophagus for resulting thermal lesions.
  Interventions: Device: Circa™ Probe

INTERVENTIONS:
Device: Circa™ Probe — The Circa™ probe will be used to monitor esophageal temperature and guide ablation power and duration during the RFCA procedure. Following ablation esophagoscopy will be performed to assess for esophageal lesions.
  Other Names: CIRCA; K112376

SUMMARY:
The purpose of this study is to determine if the use of Circa™ temperature monitoring system during ablation procedures will reduce the risk of esophageal lesions or damage. Esophageal lesions caused by ablation could later develop into a potentially fatal atrio-esophageal fistula, which is hole between the upper chamber of the heart and the esophagus. Although development of atrio-esophageal fistula following atrial fibrillation ablation is extremely rare, the complication is severe and potentially life-threatening. Therefore, monitoring of esophageal temperatures has been adopted to prevent the development of esophageal lesions. The Circa™ temperature monitoring system allows cardiac electrophysiologists to monitor and thereby limit temperatures as well as duration of ablation in the esophagus throughout the procedure.

DETAILED DESCRIPTION:
Dr. Gregory Feld, M.D. is conducting a research study to find out more about the short-term effects on the esophagus of left atrial ablation (guided by Circa™ esophageal temperature monitoring system). The financial supporter of this study is Circa Scientific, LLC.

When the investigators perform a radiofrequency catheter ablation (RFCA) at UCSD, the investigators routinely use the Circa™ temperature monitor system to prevent damage to the esophagus. For this study, patients will receive an esophagoscopy, a procedure in which a flexible tube with a camera is inserted through the mouth into the esophagus. The esophagoscopy will be conducted the next day following the ablation procedure to examine the lining of the esophagus for possible lesions or damage. Patients are asked to participate in this study because they are scheduled to have an ablation for atrial fibrillation (AF). There will be approximately 40 participants in this study at the University of California, San Diego (UCSD) Cardiovascular Center. The use of the Circa™ temperature monitoring system used in standard ablation procedures at UCSD and will be used whether or not patients decide to participate in this study. Using esophagoscopy, this study will evaluate the lining of the esophagus, or swallowing tube between the throat and stomach, the day following atrial fibrillation ablation by using an endoscope, flexible tube equipped with a camera.

Patients enrolled in the study will proceed to their standard of care ablation procedure for treatment of atrial fibrillation. There will be no changes to the ablation as part of this research study. The Circa™ temperature monitor system will be used throughout the ablation as is standard clinical care for all patients receiving AF ablations at UCSD. For research purposes only, patients will undergo an esophagoscopy, or endoscopic evaluation of the esophagus, the next day following the atrial fibrillation ablation. This procedure will take 40-45 minutes, and will involve inserting a flexible probe (tube) with a camera, into the throat and esophagus (swallowing tube), where it will be inspected for any damage (thermal lesions) caused during the ablation procedure.

Following the procedure, patients will be monitored in the usual fashion in the procedure treatment unit (PTU), as is standard of care following AF ablation. Ablation patients will be discharged from the hospital in a standard manner after esophagoscopy and asked to schedule a follow-up appointment following ablation, as is standard of care. There will not be any research follow-up for this study. If for any reason patients cannot complete the ablation or esophagoscopy procedure, patient will be withdrawn from study.

ELIGIBILITY:
Inclusion Criteria:

* Must have atrial fibrillation and be scheduled for AF ablation, during which the Circa esophageal temperature probe will be used to guide ablation.
* Must give written informed consent

Exclusion Criteria:

* Patient's refusal to participate in the study
* Any known esophageal disease or prior injury that would preclude esophagoscopy
* Any complications occuring during or after AF ablation that would result in esophagoscopy being an added significant risk to the patient beyond the known potential risks from the esophagoscopy
* Prior AF ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Feld, MD, Principal Investigator — UC San Diego
Locations (1):
- Sulpizio Cardiovascular Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinek M, Bencsik G, Aichinger J, Hassanein S, Schoefl R, Kuchinka P, Nesser HJ, Purerfellner H. Esophageal damage during radiofrequency ablation of atrial fibrillation: impact of energy settings, lesion sets, and esophageal visualization. J Cardiovasc Electrophysiol. 2009 Jul;20(7):726-33. doi: 10.1111/j.1540-8167.2008.01426.x. Epub 2009 Feb 2. PMID 19207781
- [Background] Dagres N, Anastasiou-Nana M. Prevention of atrial-esophageal fistula after catheter ablation of atrial fibrillation. Curr Opin Cardiol. 2011 Jan;26(1):1-5. doi: 10.1097/HCO.0b013e328341387d. PMID 21099683
- [Background] Halm U, Gaspar T, Zachaus M, Sack S, Arya A, Piorkowski C, Knigge I, Hindricks G, Husser D. Thermal esophageal lesions after radiofrequency catheter ablation of left atrial arrhythmias. Am J Gastroenterol. 2010 Mar;105(3):551-6. doi: 10.1038/ajg.2009.625. Epub 2009 Nov 3. PMID 19888201
- [Background] Sause A, Tutdibi O, Pomsel K, Dinh W, Futh R, Lankisch M, Glosemeyer-Allhoff T, Janssen J, Muller M. Limiting esophageal temperature in radiofrequency ablation of left atrial tachyarrhythmias results in low incidence of thermal esophageal lesions. BMC Cardiovasc Disord. 2010 Oct 26;10:52. doi: 10.1186/1471-2261-10-52. PMID 20977747
- [Background] Zellerhoff S, Ullerich H, Lenze F, Meister T, Wasmer K, Monnig G, Kobe J, Milberg P, Bittner A, Domschke W, Breithardt G, Eckardt L. Damage to the esophagus after atrial fibrillation ablation: Just the tip of the iceberg? High prevalence of mediastinal changes diagnosed by endosonography. Circ Arrhythm Electrophysiol. 2010 Apr;3(2):155-9. doi: 10.1161/CIRCEP.109.915918. Epub 2010 Mar 1. PMID 20194799
- [Background] Carroll BJ, Contreras-Valdes FM, Heist EK, Barrett CD, Danik SB, Ruskin JN, Mansour M. Multi-sensor esophageal temperature probe used during radiofrequency ablation for atrial fibrillation is associated with increased intraluminal temperature detection and increased risk of esophageal injury compared to single-sensor probe. J Cardiovasc Electrophysiol. 2013 Sep;24(9):958-64. doi: 10.1111/jce.12180. Epub 2013 Jun 7. PMID 23746064
- [Background] Feld GK, Tate C, Hsu J. Esophageal temperature monitoring during AF ablation: multi-sensor or single-sensor probe? J Cardiovasc Electrophysiol. 2013 Dec;24(12):E24. doi: 10.1111/jce.12305. Epub 2013 Nov 14. No abstract available. PMID 24118278
- [Background] ASGE Standards of Practice Committee; Evans JA, Early DS, Fukami N, Ben-Menachem T, Chandrasekhara V, Chathadi KV, Decker GA, Fanelli RD, Fisher DA, Foley KQ, Hwang JH, Jain R, Jue TL, Khan KM, Lightdale J, Malpas PM, Maple JT, Pasha SF, Saltzman JR, Sharaf RN, Shergill A, Dominitz JA, Cash BD; Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy. The role of endoscopy in Barrett's esophagus and other premalignant conditions of the esophagus. Gastrointest Endosc. 2012 Dec;76(6):1087-94. doi: 10.1016/j.gie.2012.08.004. No abstract available. PMID 23164510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Circa™ Probe
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: In two patients in each group of 20 patients originally approved by the IRB for enrollment (total 40 for the study) either the endoscopy could not be performed (2 patients) or the patients declined to undergo endoscopy after the procedure (2 patients). Thus, only 36 patients ended up completing the study and could be included in the data analysis.
Arm/Group | Circa™ Probe
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Esophageal Lesions.
Description: The number of esophageal lesions observed by esophageal endoscopy after left atrial radiofrequency catheter ablation for atrial fibrillation.
Time Frame: Day 1
Population: Among the 36 patients in this study, 18 underwent esophagoscopy immediately after ablation for atrial fibrillation and 18 underwent esophagoscopy 1 day after ablation. The pre-specified intent of this analysis was to determine the number of esophageal lesions, if any, in the entire group of 36 patients, with analysis done immediately or one day after ablation, so as to not miss any lesions which may have taken up to 24 hours to appear.
Measure: Number; unit: esophageal lesions
Groups:
- Circa™ Probe: Circa™ Probe: The Circa™ probe will be used to monitor esophageal temperature and guide ablation power and duration during the RFCA procedure. Following ablation, esophagoscopy will be performed to assess for any esophageal lesions. The first phase of the study consisted of patients who were to undergo esophagoscopy immediately after ablation and the second phase of the study in patients 24 hours after ablation.
Arm/Group | Circa™ Probe
Number analyzed (Participants) | 36
esophageal lesions | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each study participant from the time of ablation through the time of esophagoscopy, which included immediately after ablation in the first phase of the study (18 patients) and 24 hours after ablation in the second phase of the study (18 patients).
Arm/Group | Circa™ Probe
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: Part 1 (2015-03-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02467166/Prot_000.pdf
  • Study Protocol: Part 2 (2016-12-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT02467166/Prot_001.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT02467166/SAP_002.pdf